CLINICAL TRIAL: NCT00418444
Title: Randomized Control Trial of a Group Therapy Intervention Addressing Body Image and Psychosocial Functioning for Women With Breast Cancer
Brief Title: Body Image and Psychosocial Functioning in Women With Breast Cancer: Can We Fix What We've Broken?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CBCRA#017731
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2007-01

CONDITIONS: Breast Neoplasms
Keywords: Breast cancer,group psychotherapy,RCT,women's mental health
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Behavioral: Group Therapy Intervention

SUMMARY:
The purpose of this study is to test an innovative intervention geared towards issues of identity, body image and sexuality, and to examine the intervention for its impact on body image, quality of life, psychosocial/sexuality/relational functioning.

DETAILED DESCRIPTION:
Breast cancer is the most frequently diagnosed cancer in women with 1 in 10 Canadian women being diagnosed in their lifetime. There has been an increase in the number of survivors due to advances in treatment and early detection, and increased scientific attention has been focused on patients' quality of life during and after treatment. The majority of survivors do well after the initial adjustment within the first 2 years post-treatment. However, depending on when assessed after treatment completion, a wide range of cancer survivors either score at levels suggestive of a psychiatric diagnosis or are diagnosed with a psychological problem. Furthermore, a subset of survivors experience adjustment problems long after treatment completion. Approximately 20% to 40% of survivors develop sexual and body image problems following breast cancer and treatment and these difficulties tend to persist several years after treatment completion.

This study aims to test an innovative intervention geared towards issues of identity, body image and sexuality and to examine the intervention for its impact on body image and quality of life, psychosocial and sexual functioning and relational functioning.

One hundred and eighty women who have completed treatment for breast cancer will be randomized into either intervention: an 8 weekly psychosocial group support or control condition (standard care + written educational material). All subjects will be followed for 1 year post-intervention. It is hypothesized that, compared to control subjects who receive standard care and educational materials, subjects participating in an 8 weekly psychosocial group support will have higher levels of relationship support/functioning, and that the group differences will be maintained over the 1-year follow up period.

ELIGIBILITY:
Inclusion Criteria:

* women with primary breast cancer
* age between 18 and 65 years
* completed adjuvant treatments
* Stage I,II,III cancer of the breast with no metastatic disease

Exclusion Criteria:

* presence of any metastases
* history of major psychiatric disorder as defined by the DSM-IV
* inability to speak or read English for questionnaire completion
* failure to provide informed consent
* currently participating in a therapist-led psychosocial support group

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Self image and communication(using standardized instruments)

SECONDARY OUTCOMES:
Psychosocial and psychosexual functioning (using standardized instruments)
Relational functioning, quality of life and health care utilization (using standardized instruments)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jane Esplen, PhD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario

REFERENCES:
- [Derived] Esplen MJ, Wong J, Warner E, Toner B. Restoring Body Image After Cancer (ReBIC): Results of a Randomized Controlled Trial. J Clin Oncol. 2018 Mar 10;36(8):749-756. doi: 10.1200/JCO.2017.74.8244. Epub 2018 Jan 22. PMID 29356610